CLINICAL TRIAL: NCT06087705
Title: Real-life Assessment of the Safety and Performance of the SYNOVIUM HCS Device
Acronym: YNOVIUM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LCA Pharmaceutical (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: YNOVIUM
Record Dates: First submitted 2023-02-06; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Gonarthrosis
Keywords: hyaluronic acid
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Intra-articular injection of hyaluronic acid — The injection must necessarily be performed by a practitioner in compliance with the rules of asepsis.
  Procedure of use:
  * Before the injection, a rigorous prior disinfection of the area to be treated will be carried out.
  * Check the integrity of the sterility protector.
  * Take the syringe and remove the protective tip.
  * Hold the syringe body and insert a sterile intra-articular injection needle into the Luer-Lock system.
  * Gently turn the needle clockwise to secure the needle in the Luer-Lock system.
  * A visual check of the attachment of the needle will be carried out.
  * Remove the needle cap.
  * Inject slowly.

SUMMARY:
Patients who are to benefit from an injection of SYNOVIUM HCS as part of their care will be offered to participate in this study. Patients will need to sign a consent form to participate. Prior to SYNOVIUM HCS injection, patients will be asked a series of questions regarding their pain and disability. Data collected during follow-up visits can be compared to pre-injection data.

DETAILED DESCRIPTION:
Inclusion period: 6 months

Follow-up period:

* 6-month follow-up, after intra-articular injection with extension

  * 1 single syringe of SYNOVIUM HCS (3 mL),
  * Controls scheduled at 1 week, 1, 3, 6 months and up to 1 year
  * Additional control (single) in the event of leaving the study if this takes place outside the scheduled visit dates and before 1 year, for medical reasons
* Duration of the study: Overall time estimated at 18 months
* In this open-label CI, the group itself is used as a control, by comparing the scores on inclusion with those of the various control visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient with radiologically characterized gonarthrosis (stages Kellgren & Lawrence grades I to III)
* Patient with walking pain (WOMAC A1) at least equal to 2 on the Likert scale 0-4
* Patient to benefit from an injection of SYNOVIUM HCS as part of his treatment
* Patient agreeing to participate in the study
* Patient affiliated to a social security scheme or benefiting from such a scheme

Exclusion Criteria:

* Viscosupplementation less than 6 months old
* Intra-articular corticosteroid injection less than 2 months old
* Inflammatory arthritis or active infectious of the knee studied
* History of surgery of the lower limb concerned
* Kellgren & Lawrence grades not defined
* Known hypersensitivity to hyaluronic acid or chondroitin sulfate
* Pregnant or breastfeeding women
* Patient under guardianship, curatorship or judicial safeguard
* Patient participating in another clinical investigation, at the time of inclusion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
device performance | 6 months
  evolution of the pain sub-score of the WOMAC (universities of Western Ontario and McMaster) index (A). The higher the score, the more the knee osteoarthritis has a functional impact.

SECONDARY OUTCOMES:
Complication | 1 year
  complication rate
recovery of autonomy | 1 year
  Evolution of the disability according to the patient (Likert scale 0-10, higher scores mean better outcome)
Evolution of the pain | 1 year
  Evolution of the pain sub-score (WOMAC A)(universities of Western Ontario and McMaster) index (A). (Higher scores mean worse outcome)
Stiffness | 1 year
  Evolution of the stiffness sub-score (WOMAC B) (universities of Western Ontario and McMaster) index (B). (Higher scores mean worse outcome)
Function | 1 year
  Evolution of the function sub-score (WOMAC C) (universities of Western Ontario and McMaster) index (C). (Higher scores mean worse outcome)
responder patients | 1 year
  Rate of responder patients according to the OMERACT-OARSI criteria (to the treatment, in knee osteoarthritis) (0% (no responder) to 100% (all responder))
Impact of the injection on concomitant treatments | 1 year
  Recording of the consumption of analgesics and NSAIDs
long-term performance of the SYNOVIUM HCS device | 1 year
  Rate of patients having reached 1 year, without intervention on the knee concerned
Investigator's general assessment | 1 year
  General assessment by the investigator at the end of the study. (Likert scale 0-3, higher scores mean better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique BARON, Principal Investigator — CRRF en Milieu Marin de Trestel
Locations (1):
- CRRF en Milieu Marin de Trestel, Saint-Brieuc, France

IPD SHARING:
Plan to Share IPD: No